CLINICAL TRIAL: NCT03992703
Title: Clinical Impact of Rapid Susceptibility Testing on MHR-SIR Directly From Blood Cultures
Brief Title: Clinical Impact of Rapid AST Directly From Blood Cultures
Acronym: MHR-BC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MHR-BC
Record Dates: First submitted 2019-06-14; First posted 2019-06-20 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Bacterial Infections
Keywords: Clinical impact; Bacteremia; Antibiotic; Blood cultures; Enterobacteriaceae; Staphylococcus aureus
MeSH Terms: conditions — Bacterial Infections; Bacteremia; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard strategy: This group has been treated with antibiotic susceptibility testing on a conventional Mueller-Hinton medium with reading after 24 hours of incubation (Period 1: from July 1, 2015 to December 31, 2016)
- Rapid strategy: This group has been treated with antibiotic susceptibility testing on a rapid Mueller-Hinton medium after 8 hours of incubation (period 2: January 1, 2017 to June 30, 2018)

SUMMARY:
Bacteremia is defined as pathogenic bacteria presence in blood as evidenced by positive blood cultures. These bacteremia have significant consequences in terms of morbidity and mortality (ref. 1,2,3). They can lead to a state of septic shock that is life-threatening for the patient and must be treated as a matter of urgency. Any delay in treatment is detrimental to the patient. Management is based on prescription of probabilistic antibiotic therapy as soon as bacteremia is suspected.

At the Groupe Hospitalier Paris Saint Joseph (GHPSJ), as soon as a blood culture is known to be positive, the Mobile Clinical Microbiology Unit (UMMC) is notified in real time. The UMMC infectiologist, in consultation with the microbiologist, evaluates microbiological data and compares them with clinical data in order to prescribe probabilistic antibiotic therapy in the patient's bed. The possible adaptation of antibiotic treatment then depends on the results of antibiotic susceptibility test.

Early adaptation of antibiotic treatment to antibiotic susceptibility data, to reassess ineffective treatment or to reduce antibiotic therapy spectrum, significantly improves patient prognosis: it is therefore important that the laboratory makes antibiotic susceptibility test results available to the clinician as early as possible.

DETAILED DESCRIPTION:
The standard method based on diffusion on agar medium on conventional CBM allows antibiotic susceptibility results the test to be rendered within 24 hours. Many so-called rapid methods (Accelerate PhenoTM system, VITEK 2 Rapid Identification and Susceptibility Testing System,...) have been developed to improve antibiotic susceptibility testing speed from positive blood cultures. However, these approaches are costly and not exhaustive in terms of antibiotic panels tested.

The Mueller-Hinton Rapid-SIR (MHR-SIR) i2a medium has been developed. It is an agar medium allowing an early reading of antibiotic susceptibility test due to contrasting agents presence in culture medium which facilitates antibiotic susceptibility test results reading in less than 8 hours on a majority of fast-growing bacteria, in particular Enterobacteriaceae and golden staphylococci.

A prospective evaluation of the Mueller-Hinton Rapid-SIR (MHR-SIR) medium's performance directly from blood cultures was conducted in GHPSJ laboratory and published in 2018 with very satisfactory results obtained in less than 8 hours with a correlation > 97% compared to the standard MH method (Results published in DMID ref.5) at a very moderate cost of 5 euros for 16 antibiotics in free choice; The additional cost compared to the traditional MH is 20% or 0.4 euros per agar. In view of excellent results of the study, this technique has replaced the traditional MH technique in GHPSJ laboratory since January 2017, allowing UMMC to propose more quickly adaptations of probabilistic antibiotic therapy.

The use of the MHR-SIR medium has never been evaluated in a clinical context. The objective of this pioneering study is to routinely evaluate the rendering clinical impact of the rapid antibiotic susceptibility test MHR-SIR (i2a) after 8 hours of incubation directly from the blood cultures.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in a clinical department of the Groupe Hospitalier Paris Saint-Joseph
* Patient for whom a blood culture and antibiotic susceptibility test have been prescribed in the event of suspected bacteremia
* Patient with a positive blood culture with enterobacteriaceae or Gram-positive cocci suggestive of Staphylococcus sp.
* Patient whose antibiotic susceptibility test was performed on conventional Mueller-Hinton medium between July 1, 2015 and December 31, 2016 or on rapid Mueller-Hinton medium between January 1, 2017 and June 30, 2018 (date of antibiotic susceptibility test)
* Adult patient (age > 18 years)
* Patient with social care

Exclusion Criteria:

* Bacteremic patient with bacteria other than enterobacteriaceae or Gram-positive cocci suggestive of Staphylococcus sp.
* Patient objecting to use of their data for this research
* Patient under guardianship or curatorship (unless consent is provided)
* Patient deprived of liberty
* Patient under justice protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with a positive blood culture and whose antibiotic susceptibility test was performed on conventional Mueller-Hinton medium between July 1, 2015 and June 30, 2018
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Differences in average time between the prescribing physician's request for examination and the first change in prescribed probabilistic antibiotic therapy following the rendering of results between two groups of patients. | 6 months
  Differences in average time between the prescribing physician's request for examination and the first change in prescribed probabilistic antibiotic therapy following the rendering of results between
  * a "standard strategy" group that has been treated with antibiotic susceptibility testing on a conventional Mueller-Hinton medium with reading after 24 hours of incubation (Period 1: from July 1, 2015 to December 31, 2016);
  * a "rapid strategy" group that has been treated with antibiotic susceptibility testing on a rapid Mueller-Hinton medium after 8 hours of incubation (period 2: January 1, 2017 to June 30, 2018).
  Prescribing changes taken into account include the introduction of an antibiotic, a change in the prescribed antibiotic or a change in its dosage (escalation, de-escalation).

SECONDARY OUTCOMES:
Percentage of patients with escalation and de-escalation of prescribed probabilistic antibiotic therapy | 6 months
  Evaluate the rendering impact of a rapid antibiotic susceptibility testing (8 hours) in bacteriemic patients compared to standard antibiotic susceptibility testing (24 hours) on escalation and de-escalation of prescribed probabilistic antibiotic therapy by percentage, after rendered results.
Average number of days of broad-spectrum antibiotic therapy | 6 months
  Evaluate the rendering impact of a rapid antibiotic susceptibility testing (8 hours) in bacteriemic patients compared to standard antibiotic susceptibility testing (24 hours) on prescribing broad-spectrum antibiotic therapy by calculating average number of days for both groups.
Average oral relay time for antibiotics | 6 months
  Evaluate the rendering impact of a rapid antibiotic susceptibility testing (8 hours) in bacteriemic patients compared to standard antibiotic susceptibility testing (24 hours) on antibiotics oral relay by calculating the average oral relay time for both groups.
Intra-hospital mortality prevalence of infectious origin | 6 months
  Evaluate the rendering impact of a rapid antibiotic susceptibility testing (8 hours) in bacteriemic patients compared to standard antibiotic susceptibility testing (24 hours) on in-hospital mortality of infectious origin.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude NGUYEN VAN, Doctor, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perillaud C, Pilmis B, Diep J, Pean de Ponfilly G, Vidal B, Couzigou C, Mizrahi A, Lourtet-Hascoet J, Le Monnier A, Nguyen Van JC. Prospective evaluation of rapid antimicrobial susceptibility testing by disk diffusion on Mueller-Hinton rapid-SIR directly on blood cultures. Diagn Microbiol Infect Dis. 2019 Jan;93(1):14-21. doi: 10.1016/j.diagmicrobio.2018.07.016. Epub 2018 Jul 31. PMID 30149988
- [Background] Garnacho-Montero J, Gutierrez-Pizarraya A, Escoresca-Ortega A, Fernandez-Delgado E, Lopez-Sanchez JM. Adequate antibiotic therapy prior to ICU admission in patients with severe sepsis and septic shock reduces hospital mortality. Crit Care. 2015 Aug 27;19(1):302. doi: 10.1186/s13054-015-1000-z. PMID 26307060
- [Background] Brun-Buisson C, Doyon F, Carlet J, Dellamonica P, Gouin F, Lepoutre A, Mercier JC, Offenstadt G, Regnier B. Incidence, risk factors, and outcome of severe sepsis and septic shock in adults. A multicenter prospective study in intensive care units. French ICU Group for Severe Sepsis. JAMA. 1995 Sep 27;274(12):968-74. PMID 7674528
- [Background] Ferrer R, Martin-Loeches I, Phillips G, Osborn TM, Townsend S, Dellinger RP, Artigas A, Schorr C, Levy MM. Empiric antibiotic treatment reduces mortality in severe sepsis and septic shock from the first hour: results from a guideline-based performance improvement program. Crit Care Med. 2014 Aug;42(8):1749-55. doi: 10.1097/CCM.0000000000000330. PMID 24717459
- See also: Pubmed — https://www.ncbi.nlm.nih.gov/pubmed/30149988